CLINICAL TRIAL: NCT02921828
Title: Pomalyst®Capsules Special Use-results Surveillance (All-case Surveillance)
Brief Title: A Safety and Efficacy of Pomalyst® Capsules Under the Actual Use in All Patients Who Are Treated With Pomalyst at a Dose of 1 mg, 2 mg, 3 mg, or 4 mg
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-Celgene-JP-PMS-002
Record Dates: First submitted 2016-09-30; First posted 2016-10-03 (Estimated); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Multiple Myeloma
Keywords: Pomalyst; Teratogenicity; bone marrow suppression; thromboembolism; peripheral neuropathy; infection; tumour lysis syndrome; somnolence; depressed level of consciousness; confusion; fatigue; dizziness; acute renal failure; heart failure; arrhythmia; interstitial pneumonia; hypersensitivity; hepatic function disorder; jaundice
MeSH Terms: conditions — Multiple Myeloma; Teratogenesis; Thromboembolism; Peripheral Nervous System Diseases; Infections; Tumor Lysis Syndrome; Sleepiness; Consciousness Disorders; Confusion; Fatigue; Dizziness; Acute Kidney Injury; Heart Failure; Arrhythmias, Cardiac; Lung Diseases, Interstitial; Hypersensitivity; Liver Diseases; Jaundice

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Multiple myeloma patients who received Pomalyst: Among relapsed or refractory multiple myeloma patients, all patients who received Pomalyst will be targeted in this surveillance.

SUMMARY:
1. Planned enrollment period One year (The planned number of patients to be enrolled is set to 400 patients.) Since all patients who are prescribed with Pomalyst are registered in RevMate®, enrollment using the Registration Form of the surveillance will be completed at the time when the planned number of patients to be enrolled is reached. During a period until conditions for approval are removed, a system enabling to retrospectively collect appropriate information based on patient data from RevMate® will be, as necessary, maintained.
2. Planned duration of the surveillance Anticipated to be 2 years and 6 months from the start date of release of Pomalyst

ELIGIBILITY:
Inclusion Criteria:

* Among relapsed or refractory multiple myeloma patients, all patients who received Pomalyst will be targeted in this surveillance.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among relapsed or refractory multiple myeloma patients, all patients who received Pomalyst will be targeted in this surveillance.
Sampling Method: Non-Probability Sample
Enrollment: 1149 (Actual)
Dates: Start 2015-04-30 (Actual); Primary Completion 2015-12-10 (Actual); Study Completion 2015-12-10 (Actual)

PRIMARY OUTCOMES:
Adverse event (AE) | 3 years
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Jinshu Cho, Study Director — Celgene
Locations (2):
- Local Institution - Japan, No City Provided, New Jersey, United States
- Shinko Hospital, Kobe, Hyōgo, Japan